CLINICAL TRIAL: NCT02623530
Title: The Teaching of Critical Thinking for Nursing Students: A Randomized Controlled Pilot Study
Brief Title: Critical Thinking in Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Fábio da Costa Carbogim, Phd student, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 1.274.735; 45536215.9.0000.5392 (Other: USaoPaulo)
Record Dates: First submitted 2015-12-01; First posted 2015-12-07 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Thinking
Keywords: Nursing; Nursing education research; Critical thinking; Decision Making
MeSH Terms: interventions — Early Intervention, Educational

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (Active Comparator): Control group: to implement educational intervention focusing on first aid for developing critical thinking (CT) skills and disposition, through the Problem Based Learning (PBL), not based on the Active Learning Model for Critical Thinking (MEAPC).
  Interventions: Other: Educational intervention
- Experimental group (Experimental): Experimental group: to implement educational intervention focusing on first aid for developing critical thinking (CT) skills and disposition, through the Problem Based Learning (PBL), based on the Active Learning Model for Critical Thinking (MEAPC).
  Interventions: Other: Educational intervention

INTERVENTIONS:
Other: Educational intervention — Control Group: An educational intervention focusing on first aid for the development of skills and dispositions of critical thinking. For this group will be taught the contents of first aid through the Methodology of PBL without the support MEAPC.
  Experimental Group: An educational intervention focusing on first aid for the development of skills and dispositions of critical thinking. For this group will be taught the contents of first aid through Methodology PBL, supported by the MEAPC.

SUMMARY:
Considering the need for an intervention in the context of the Brazilian nursing education, in order to develop the skills and dispositions for critical thinking (CT), this study aims to fill this gap through a first aid course, comparing a group control and an experimental group. In this study will be used two tests, California Critical Thinking Dispositions Inventory (CCTID) to review arrangements for the CT, and California Critical Thinking Skills Test (CCTST) to evaluate CT skills, both marketed (Facione N, Facione PA, 2009 , 2011). Therefore, in order to facilitate the assimilation of PC skills during the course, we prepared the model of Active Teaching for Critical Thinking (MEAPC): characterized by a teaching method proposed by the author of this work, who understands the educational activity active and intentional as mobilizing higher mental processes fundamental to the development of the CT.

DETAILED DESCRIPTION:
In Brazil there are few studies produced about Critical Thinking (CT), and the field of Brazilian nursing are unknown type of intervention research to assess / provisions initially measure and skills development / PC skills. Thus, the research question to be answered is: Students undergo an educational intervention focused on first aid care based on the Problem Based Learning (PBL) and guided by Active Teaching Model for Critical Thinking (MEAPC), have better results for PC skills and provisions compared to students learning the same content from PBL without MEAPC?

* STUDY OBJECTIVES

General Purpose:

Create, implement and evaluate an educational intervention for nursing students focusing on first aid, to develop skills and PC provisions, based on Problem Based Learning (PBL) and guided by Active Teaching Model for Critical Thinking (MEAPC) .

Specific Objectives:

* Create an educational intervention focusing on first aid, to develop skills and PC provisions, through the PBL, guided by MEAPC (experimental group) and with PBL and without MEAPC (control group);
* Apply the educational intervention focusing on first aid for the development of skills and PC provisions, through the PBL, guided by MEAPC (experimental group) and the PBL and without MEAPC (control group);
* Evaluate the experimental group and control (before and immediately after the intervention) PC skills and dispositions, respectively, through the test California Critical Thinking Disposition Inventory (CCTDI) and California Critical Thinking Skills Test (CCTST);
* Compare possible differences between the two groups of students (experiment and control) in relation to age and sex;
* Evaluate the effectiveness of MEAPC associated with PBL, comparing the performance of the experimental group and control;
* Assess the educational intervention through knowledge of students using tests ten true and false statements (T or F test) applied before and immediately after the intervention.

STUDY ASSUMPTIONS

This study will be developed based on five assumptions, explained below:

* Students who participate in the educational intervention focused on first aid care, based on the PBL-driven MEAPC will get better results in the test California Critical Thinking Dispositions Inventory (CCTID) and test California Critical Thinking Skills Test (CCTST), which students attending the educational intervention aimed at answering first aid, based on the PBL, but not being guided by MEAPC;
* Older students (22 and older) will get better results in the tests California Critical Thinking Dispositions Inventory (CCTID) and California Critical Thinking Skills Test (CCTST) than younger students (under 22 years) in the experiment and control groups;
* There will be no significant differences regarding gender in relation to tests California Critical Thinking Dispositions Inventory (CCTID) and California Critical Thinking Skills Test (CCTST) compared the experimental and control groups;
* The evaluation of educational intervention through knowledge of students using true and false statements test (V or F) applied before and immediately after the intervention, developed quantitative improvement in results.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate nursing students who are enrolled from first to third year;
* Undergraduate nursing students who agreed to participate in the study by signing the free and informed consent;
* Undergraduate nursing students residing in the Zona da Mata of Minas Gerais, Brazil.

Exclusion Criteria:

* Undergraduate nursing students who are not enrolled from first to third year;
* Undergraduate nursing students who does not agreed to participate in the study by signing the free and informed consent.
* Undergraduate nursing students who does not residing in the Zona da Mata of Minas Gerais, Brazil.

Ages: 17 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 102 (Actual)
Dates: Start 2015-10; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
California Critical Thinking Skills Test (CCTST) | one year
  It is now considered the main test for measurement of critical thinking skills. The test is divided into ranges that represent the skills of critical thinking, analysis, evaluation, inference, deduction, induction and general reasoning skills. The test has 34 questions (about five questions to assess each critical thinking skill) with four possible answers listed from A to D. Students must choose only one answer that they consider relevant to the question asked. The test filling time takes around 50 minutes.
California Critical Thinking Dispositions Inventory (CCTID) | one year
  Have your items divided into seven scales that represent attitudes of the critical thinker: seeking the truth, open mind, analyticity, systematic, self-confidence, curiosity and cognitive maturity. The test has 75 assertions (about 11 for each assertive attitude) from which students must indicate their level of agreement or disagreement on a Likert scale of six points. The test filling time takes around 15 to 20 minutes.

SECONDARY OUTCOMES:
Evaluation of educational intervention | one year
  The evaluation of educational intervention through knowledge of students using true and false statements test (V test or F).

CONTACTS AND LOCATIONS:
Overall Officials: Vilanice F Püschel, Phd, Study Director — University of Sao Paulo
Locations (1):
- Universidade Federal de Viçosa, Viçosa, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
Data will be analyzed until June 2016, and subsequently arranged for publication.